CLINICAL TRIAL: NCT05362500
Title: Comparative Study Between Chemical Peeling With 70% Glycolic Acid and Intradermal Transamine for the Treatment of Melasma.
Brief Title: Comparison of Chemical Peeling Agent With Transamine for Treatment of Melasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Naheed khan, principal investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHatd-ETH-22-derm-22; 131/CPSP (Other: CPSP)
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid; Tranylcypromine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A 70% Glycolic acid (Active Comparator): Group A: contain 27 patients which had been treated every 2 weeks for 12 weeks with 70% glycolic acid to assess chemical peeling and cold water was used for washing to stop peeling
  Interventions: Drug: Glycolic Acid 70%
- Group B intradermal tranexamic acid (Active Comparator): Group B: contain 27 patients treated with an intradermal injection of 0.05 mL of tranexamic acid solution in normal saline (4 mg/mL) into the melasma lesion at 1 cm distance using a sterile insulin syringe, weekly for 12 weeks
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Glycolic Acid 70% — Group A: contain 27 patients which had been treated every 2 weeks for 12 weeks with 70% glycolic acid to assess chemical peeling and cold water was used for washing
  Other Names: Peeling agent
  Arms: Group A 70% Glycolic acid
Drug: Tranexamic acid injection — Group B: contain 27 patients treated with an intradermal injection of 0.05 mL of tranexamic acid solution in normal saline (4 mg/mL) into the melasma lesion at 1 cm distance using a sterile insulin syringe, weekly for 12 weeks
  Other Names: transamine injection
  Arms: Group B intradermal tranexamic acid

SUMMARY:
Melasma is an acquired skin disorder characterized by hyper-melanosis. Melasma is a term that originates from the Greek root "melas" (black color) and was formerly known as chloasma. Melasma is more common in sun-exposed tissues such as the cheeks, chin, upper lip, and forehead. Melasma is a common dermatological disorder with a frequency of 8.8 percent in the United States, but it can be as high as 40 percent amongst females. Melasma affects mostly ladies and is most common throughout their reproductive years .

Melasma causes an increase in melanin pigment synthesis owing to a surge in the number of melanosomes, which are membrane-bound cell organelles inside melanocytes where melanin biosynthesis occurs and is transported to keratinocytes. Except in rare situations, the number of melanocytes will not be enhanced. Melanocytes will grow in size, and dendrites will become more visible. Despite the fact that the specific causation is unknown, some elements are thought to have a role in the pathophysiological mechanisms of melasma). Among these, sun exposure (UV light) is the most powerful primary trigger for its growth, which explains melisma's propensity for certain areas of the body. Other major determinants include genetic predisposition, and female hormones - both endogenous (that is, during pregnancy) and exogenous (that is, during pregnancy) (contraceptives and hormone replacement therapy). Thyroid problems, medications, and cosmetics can all be aggravating factors. Evaluation and prevention of triggering variables are essential in order to avoid recurrence .

The peeling effect of glycolic acid is due to chemo exfoliation capabilities, that rely upon aiding the elimination of keratinocytes, resulting in melanin reduction and speeding up the regeneration of skin. TA suppresses UV-stimulated plasmin action in keratin cells by blocking plasminogen appending to the keratin cells, resulting from lower free arachidonic acid levels or to reduced capacity of prostaglandins production, which reduces melanocyte tyrosinase activity .

The study's implications are to analyze the efficacy of these two drugs in order to assess the better outcome of patients with evidence-based management.

DETAILED DESCRIPTION:
A randomized controlled trial study (single-blind) was done In the Dermatology Unit of the CMH, Abbottabad from June to November 2021 after Ethical Review Board approval, the 54 patients aged 20-50 years after informed consent were enrolled using a technique of non-probability consecutive sampling. The sample size was determined using the WHO sample size calculator, With a significance level of 95%, power of study 80%, the ratio of sample size B: A of 1 and Assumed MASI score in Group A (Tranexamic Acid) Mean + SD = 9.37 ± 2.18, in Group B (Glycolic Acid 70%) Mean + SD = 10.25 ± 2.93. Thus, the required sample size was 54 (27 in each group).

For randomization, the final recruited 54 participants (38 females, 16 males; aged 20-50 years), recruited into two groups i.e. Group A: contain 27 patients which had been treated every 2 weeks for 12 weeks with 70% glycolic acid to assess chemical peeling and cold water was used for washing to stop peeling as displayed and Group B: contain 27 patients treated with an intradermal injection of 0.05 mL of tranexamic acid solution in normal saline (4 mg/mL) into the melasma lesion at 1 cm distance using a sterile insulin syringe, weekly for 12 weeks .

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from Melasma who attended the Dermatology department

Exclusion Criteria:

* history of hormone therapy and contraceptive pills (within the previous 12 months)
* bleeding problems or concurrent use of anticoagulants
* Topical treatment such as hydroquinone (one month prior to the research)
* Active herpes simplex, face warts or active dermatoses
* History of hypersensitivity to some of the study's components
* Pregnant or lactating females
* Patients with unrealistic expectations

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of 70%glycolic acid and intradermal transamine for treatment of melasma as assessed by MODIFIED MELASMA SEVERITY INDEX (mMASI) | 12 weeks
  Modified melasma severity index was used to measure effectiveness of both drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Naheed Khan, Principal Investigator — Cpsp
Locations (1):
- Combined military hospital, Abbottābād, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No